CLINICAL TRIAL: NCT00383578
Title: A Multicenter, Randomized, Double-Blind, Active Controlled Study to Compare the Effect of 24 Weeks Treatment With Vildagliptin 100 mg qd or Metformin 1500 mg Daily in Elderly Drug Naive Patients With Type 2 Diabetes
Brief Title: Efficacy and Safety of Vildagliptin Compared to Metformin in Elderly Drug Naive Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A2398
Record Dates: First submitted 2006-09-29; First posted 2006-10-03 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2013-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; vildagliptin; hemoglobin A1c; metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Vildagliptin (Experimental)
  Interventions: Drug: Vildagliptin 100 mg qd
- Metformin (Active Comparator)
  Interventions: Drug: Metformin 1500 mg daily

INTERVENTIONS:
Drug: Vildagliptin 100 mg qd
  Arms: Vildagliptin
Drug: Metformin 1500 mg daily
  Arms: Metformin

SUMMARY:
This study is designed to demonstrate the efficacy and safety of vildagliptin compared to metformin in elderly drug naive patients with type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* Age from 65 years to the upper age limit recommended by local prescribing information for metformin
* Drug naive patients with type 2 diabetes.
* Body mass index (BMI) in the range of 22-40 kg/m2.
* HbA1c in the range of 7 to 9% inclusive
* FPG <270 mg/dL (15 mmol/L)

Exclusion Criteria:

* A history of type 1 diabetes
* Evidence of significant diabetic complications
* Treatment with insulin or any other oral antidiabetic agents

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 335 (Actual)
Dates: Start 2006-09; Primary Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c | after 24 weeks of treatment

SECONDARY OUTCOMES:
Adverse event profile | after 24 weeks of treatment
Gastrointestinal tolerability | after 24 weeks of treatment
Patients with endpoint HbA1c <7% and patients with reduction in HbA1c > 0.7% | after 24 weeks of treatment
Change from baseline in fasting plasma glucose | after 24 weeks of treatment
Change from baseline in body weight | after 24 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Investigative Centers, Nuremberg, Germany
- Novartis Pharmaceuticals, Basel, Switzerland

REFERENCES:
- See also: Resutls for CLAF237A2398 on the Novartis clinical trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2652